CLINICAL TRIAL: NCT01733888
Title: Evaluating the Effect of Resin Infiltration and Resin Infiltration With Bleaching in Improving the Esthetics for Non Pitted Fluorosis Stains in Indian Population
Brief Title: Resin Infiltration and Resin Infiltration With Bleaching in Improving the Esthetics for Fluorosis Stains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLUORIC
Record Dates: First submitted 2012-11-14; First posted 2012-11-27 (Estimated); Results first posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Caries Infiltration; Fluorosis; Dental Care
Keywords: caries; caries infiltration; fluorosis treatment
MeSH Terms: conditions — Fluoride Poisoning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Office Bleaching (Active Comparator): Fluorosed teeth will be bleached using 35 % Hydrogen Peroxide (Pola Office, SDI, Australia) according to manufactures´ instruction.
  Interventions: Device: Office Bleaching
- Resin Infiltration (Experimental): White spots in fluorosed teeth will be infiltrated using the resin infiltrant "Icon" (DMG, Hamburg, Germany) according to manufactures´ instructions.
  Interventions: Device: Resin Infiltration
- Resin Infiltration twice (Experimental): White spots in fluorosed teeth will be infiltrated using the resin infiltrant Icon (DMG, Hamburg, Germany) according to manufactures´ instructions. Here, the infiltrant "Icon" is applied twice.
  Interventions: Device: Resin Infiltration twice
- Office Bleaching + Resin Infiltration (Experimental): Fluorosed teeth will be bleached using 35 % Hydrogen Peroxide (Pola Office, SDI, Australia). After a 20 day wash over period, these teeth will be treated with the resin infiltration intervention (Icon, DMG, Hamburg, Germany).
  Interventions: Device: Bleaching + Resin Infiltration

INTERVENTIONS:
Device: Office Bleaching — Teeth will be cleaned with pumice first, followed by placing cheek retractors and covering of the lip surface with petroleum gel. Thereafter, teeth will be dried and gingival barrier will be applied to both arches - slightly overlapping enamel and interproximal spaces. Light curing of the gingival barrier will be done in a fanning motion for 10-20 seconds. This is followed by homogeneous mixing of the powder and liquid in a powder pot the application of a thick layer of the resulting gel to all teeth undergoing treatment (35 % Hydrogen Peroxide, Pola Office, SDI, Australia). The gel will be left in place for 8 minutes and subsequently removed using a surgical aspirator tip.
  Other Names: 35 % Hydrogen Peroxide, Pola Office, SDI, Australia
  Arms: Office Bleaching
Device: Resin Infiltration — Fluorosed teeth will be isolated using a rubber dam and the resin infiltrant (Icon, DMG, Hamburg, Germany) will be applied as per manufactures' instructions. In short, tooth surface will be dried using cotton rolls and air syringe. This is followed by an etching (Icon Etch) and drying step (Icon-Dry) to open the lesion surface. Resin infiltrant will then be applied and allowed to seep in for 3 minutes followed by light curing for 40 seconds and subsequent cleaning of the surface with pumice and rubber polishing cup as well as rinsing with water for 30 sec.
  Other Names: Icon, Kit for caries infiltration, DMG, Hamburg, Germany
  Arms: Resin Infiltration
Device: Resin Infiltration twice — The intervention will be done similar to the "Resin infiltration" arm, which the exception that the icon infiltration step will be done twice.
  Other Names: Icon Kit for caries infiltration, DMG, Hamburg, Germany
  Arms: Resin Infiltration twice
Device: Bleaching + Resin Infiltration — In this arm, the fluorosed teeth of the patients will first be bleached using 35 % Hydrogen Peroxide (Pola Office, SDI, Australia) as explained in the intervention arm "Office bleaching"; followed by wash over period of 20 days. After these 20 days, patients will be recalled and the fluorosed teeth will treated according to the description in the "Resin infiltrant" intervention arm using the resin infiltrant (Icon, DMG, Hamburg, Germany) as per manufactures' instructions.
  Other Names: Icon Kit for Caries Infiltration, DMG, Hamburg, Germany; 35 % Hydrogen Peroxide, Pola Office, SDI, Australia
  Arms: Office Bleaching + Resin Infiltration

SUMMARY:
Dental fluorosis is a clinical manifestation of chronic exposure to high intakes of fluoride during the tooth development.

The present study is planned to evaluate the efficacy of Resin Infiltration technique in improving the esthetics of non-pitted fluorosis stains on permanent anterior teeth. Resin infiltration is a novel method that has shown its efficacy in improving the esthetics of various types of white spot lesions (WSLs), particularly post orthodontics WSLs, in in-situ and in-vivo studies. The Resin Infiltration technique is also known to stop the progression of caries in non cavitated lesions in both, smooth surface and interproximal lesions.

Therefore, the following trial will be conducted to assess the esthetic improvement of fluorosed permanent anterior teeth after resin infiltration and compare it with standard bleaching procedure and a combination of bleaching and Resin infiltration therapy in children with fluorosed teeth.

ELIGIBILITY:
Inclusion Criteria:

* Only the non-pitted Fluorosis opacities shall be included for this purpose; opacities in anterior teeth shall be classified according to Russell's criteria for differentiating fluoride and non- fluoride opacities
* Subjects classified /Teeth classified with dental fluorosis of 1-4 according to Thylstrup, Fejerskov classification of dental fluorosis 20
* Patients who will be willing to participate in the study and who will be accepting for recall visit.

Exclusion Criteria:

* History of allergy towards any dental material.
* Teeth classified as non-fluoride opacities
* Subjects with any systemic and local conditions not permitting the treatment
* Subjects who had undergone any treatment for dental fluorosis earlier
* Subjects with direct or indirect restorations in maxillary central or lateral incisors.
* Subjects not willing to participate in the study
* Subjects with fractured teeth maxillary central or lateral incisors.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Gugunani, Prof. Dr., Principal Investigator — Department of Pediatric and Preventive Dentistry DAV Dental College Yamuna Nagar 135001 Haryana India
Locations (2):
- India (2):
  - Department of Pediatric and Preventive Dentistry DAV Dental College, Yamuna Nagar, Haryana
  - Department of Pediatric and Preventive Dentistry DRIDS Dental College, Farīdkot, Punjab

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gugnani N, Pandit IK, Gupta M, Gugnani S, Soni S, Goyal V. Comparative evaluation of esthetic changes in nonpitted fluorosis stains when treated with resin infiltration, in-office bleaching, and combination therapies. J Esthet Restor Dent. 2017 Sep;29(5):317-324. doi: 10.1111/jerd.12312. Epub 2017 Jun 27. PMID 28654721

RESULTS

PARTICIPANT FLOW:
Groups:
- In-office Bleaching: In-office bleaching of fluorosed teeth with 35 % hydrogen peroxide (Pola Office, SDI, Australia) according to manufactures´ instruction.
- Resin Infiltration: Resin infiltration of white spots in fluorosed teeth using Icon (DMG, Hamburg, Germany) according to manufactures´ instructions.
- Resin Infiltration Twice: Resin infiltration of white spots in fluorosed teeth using Icon (DMG, Hamburg, Germany) according to manufactures´ instructions. The infiltrant "Icon" is applied twice.
- In-office Bleaching + Resin Infiltration: In-office bleaching of fluorosed teeth with 35 % hydrogen peroxide (Pola Office, SDI, Australia) according to manufactures´ instruction. After a 20 day washout period, the white spots in these teeth will be treated with resin infiltration intervention (Icon, DMG, Hamburg, Germany).
Period: Overall Study
Arm/Group | In-office Bleaching | Resin Infiltration | Resin Infiltration Twice | In-office Bleaching + Resin Infiltration
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with non-pitted fluorosis were selected from a high fluoride belt.
Groups:
- Total: Total of all reporting groups
Arm/Group | In-office Bleaching | Resin Infiltration | Resin Infiltration Twice | In-office Bleaching + Resin Infiltration | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (0.5) | 11.1 (0.9) | 11.6 (0.5) | 11.1 (0.8) | 11.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 7 | 7 | 38
  Male | 5 | 11 | 13 | 13 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hindu | 2 | 4 | 2 | 3 | 11
  Sikh | 18 | 16 | 18 | 17 | 69
Region of Enrollment [Number; unit: participants]
  India | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Esthetic Changes
Description: Pre-operative and immediate post-operative digital images are taken. These images are evaluated by two blinded evaluators using a VAS scale ranging from 1 to 7, with "1 = no improvement" and "7 = exceptional improvement".
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-office Bleaching | Resin Infiltration | Resin Infiltration Twice | In-office Bleaching + Resin Infiltration
Number analyzed (Participants) | 20 | 20 | 20 | 20
score on a scale | 1.90 (0.95) | 5.50 (1.00) | 5.53 (1.97) | 5.35 (1.21)

2. Secondary Outcome: Improvement in Brown Stains/ Change in White Opacities
Description: as for outcome 1
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-office Bleaching | Resin Infiltration | Resin Infiltration Twice | In-office Bleaching + Resin Infiltration
Number analyzed (Participants) | 20 | 20 | 20 | 20
score on a scale | 1.53 (1.07) | 4.98 (0.98) | 5.18 (1.29) | 4.40 (1.59)

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | In-office Bleaching | Resin Infiltration | Resin Infiltration Twice | In-office Bleaching + Resin Infiltration
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No